CLINICAL TRIAL: NCT05985434
Title: Prospective Observational Study on Patients Treated for Vertebral Metastasis and Vertebral Localizations of Lymphoproliferative Disease: Impact of the Treatment on the Quality of Life.
Brief Title: Prospective Observational Study on Vertebral Metastasis
Acronym: CVODMetsVert
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0009120
Record Dates: First submitted 2019-01-08; First posted 2023-08-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Vertebral Metastasis
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical treatment — decompression with or without stabilization; stabilization only; debulking; en bloc resection

SUMMARY:
Perspective observational cohort study in which the data relating to patients affected by one or more vertebral metastases or by vertebral localization of hemolifoproliferative malact and surgical treatment candidates will be collected, which will be recruited at the Complex Structure of Spine Surgery for Oncological and Degenerative Rizzoli Orthopedic Institute starting from the date of approval of the same study.

Patients of both sexes and aged 18 years or older will be included. Patients with primary (benign or malignant) tumors of the vertebrae and patients unable to consent to the study will be excluded from the study.

For each patient, in addition to the demographic data, preoperative information will be collected: type of tumor, involved vertebral levels, presence of pathological fracture, presence of visceral metastases, presence and number of other bone metastases, neurological picture according to Frankel's scale, evaluated pain according to the Visual Analogue Scale (VAS), functional status according to Karnofsky, EuroQoL-5D and SF-36 questionnaires on the quality of life; information related to the intervention itself: access, type of surgical treatment, possible preoperative embolization; intraoperative complications; information at discharge: postoperative complications, pain, neurological picture, functional status; follow-up data: pain, neurological picture, functional status, SF-36 questionnaire, late complications, local recurrence; systemic progression of the disease.

Follow-up checks will be performed at 3 months, 6 months, 12 months, 18 months, 24 and 36 months. The timing of the controls and the examinations requested by the patients will be those of normal clinical practice.

Primary endpoint is the change in quality of life (measured by scores EQ-5D and SF-36) and pain (measured using the VAS score) following surgery compared to pre-operative values.

DETAILED DESCRIPTION:
STUDY DESIGN Analytical Prospective Longitudinal cohort Not checked

RATIONALE OF THE STUDY The improvement of the systemic control of oncological diseases achieved in recent years has led to a considerable increase in patient survival; it was associated with a parallel increase in the onset of symptomatic vertebral metastases.

Such metastases are often associated with pain, mechanical instability of the spine, and even possible neurological deficits, which negatively affect the patient's quality of life and indirectly also on his survival.

The treatment of these metastases is defined by a multidisciplinary approach; surgery is indicated in the presence of mechanical instability, signs of neurological compression, intractable pain, progression of disease during systemic treatment.

The indication and the type of intervention are defined following a reference algorithm (A. Gasbarrini, M. Cappuccio, L. Mirabile, S. Bandiera, S. Terzi, G. Barbanti Bròdano, S. Boriani.) Spinal Metastases: treatment evaluation algorithm Eur Eur Med Pharmacol Sci 2004; 8: 265-274), in collaboration with the team of specialists involved.

Within the multidisciplinary team it is usually the Oncologist who provides an estimate of the prognosis quoad vitam, based on the general status of the patient and the residual therapeutic possibilities.

The goal of surgery is the local control of the disease and the improvement of the patient's quality of life.

Although there are works in the literature that demonstrate the effectiveness of surgical treatment in vertebral metastases, there are few prospective studies in which, in addition to survival, the improvement in the quality of life after the intervention is evaluated, and the improvement over time is maintained.

DESCRIPTION OF THE STUDY The study is monocentric, of a prospective observational type, with a single arm.

The study will collect data relating to patients affected by one or more vertebral metastases or by vertebral localization of hemolymphoproliferative disease candidates for surgical treatment, which will be recruited at the Complex Structure of Spine Surgery for Oncological and Degenerative Address of the Rizzoli Orthopedic Institute starting from date of approval of the study itself.

Patients of both sexes and aged 18 years or older will be included

DATA COLLECTION

For each patient will be collected, in addition to demographic data:

* preoperative information: type of tumor, vertebral levels involved, presence of pathological fracture, presence of visceral metastases, presence and number of other bone metastases, functional status according to Karnofsky (Annex 1), neurological picture according to Frankel's scale (Annex 2) , pain assessed according to the Visual Analogue Scale (VAS), EuroQoL-5D and SF-36 questionnaires on the quality of life;
* information on the intervention: access, type of surgical treatment, possible preoperative embolization; intraoperative complications;
* information at discharge: postoperative complications, pain, neurological picture, functional status;
* follow-up data: pain (VAS scale), neurological picture (according to the Frankel scale), functional status according to Karnofsky, EuroQoL-5D and SF-36 questionnaires on quality of life, late complications, local recurrence; systemic progression of the disease.

The clinical data necessary for the research will be extracted from the patient's medical record and from its source documents.

A specific data collection form will be used to collect the clinical information and the results of the analysis foreseen by the study.

For each patient included in the study, the data collection form (Case Report Form - CRF) will be compiled.

Follow-up checks will be performed, as per clinical practice, at 3 months, 6 months, 12 months, 18 months, 24 months and 36 months.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are candidates for surgery at the level of the spine at the SC of Spine Surgery, for: or vertebral metastases or or vertebral localizations from hemolymphoproliferative diseases

* Patients aged ≥ 18 years
* Patients giving written informed consent to the study

Exclusion Criteria:

* Patients with malignant or benign vertebral tumors
* Patients suffering from vertebral metastases or vertebral localizations from hemolymphoproliferative diseases for which there are no indications for surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by vertebral metastasis eligible for surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | At baseline (day 0)
  Visual Analogue Scale (VAS) patient-administered questionnaire
Pain evaluation | At 3 months follow up
  Visual Analogue Scale (VAS) patient-administered questionnaire
Pain evaluation | At 6 months follow up
  Visual Analogue Scale (VAS) patient-administered questionnaire
Pain evaluation | At 12 months follow up
  Visual Analogue Scale (VAS) patient-administered questionnaire
Pain evaluation | At 18 months follow up
  Visual Analogue Scale (VAS) patient-administered questionnaire
Pain evaluation | At 24 months follow up
  Visual Analogue Scale (VAS) patient-administered questionnaire
Pain evaluation | At 36 months follow up
  Visual Analogue Scale (VAS) patient-administered questionnaire
Quality of life evaluation | At baseline (day 0)
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Quality of life evaluation | At 3 months follow up
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Quality of life evaluation | At 6 months follow up
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Quality of life evaluation | At 12 months follow up
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Quality of life evaluation | At 18 months follow up
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Quality of life evaluation | At 24 months follow up
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Quality of life evaluation | At 36 months follow up
  EuroQoL- 5D (EQ-5D) patient-administered questionnaire
Health survey | At baseline (day 0)
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire
Health survey | At 3 months follow up
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire
Health survey | At 6 months follow up
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire
Health survey | At 12 months follow up
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire
Health survey | At 18 months follow up
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire
Health survey | At 24 months follow up
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire
Health survey | At 36 months follow up
  Short Form Health Survey 36 (SF-36) patient-administered questionnaire

SECONDARY OUTCOMES:
Prognostic factor- 1 | 3 months follow up
  Surgery-related adverse events collected by SAVES-v.2 system
Prognostic factor- 2 | 3 months follow up
  Survival rate
Prognostic factor- 1 | 6 months follow up
  Surgery-related adverse events collected by SAVES-v.2 system
Prognostic factor- 2 | 6 months follow up
  Survival rate
Prognostic factor- 1 | 12 months follow up
  Surgery-related adverse events collected by SAVES-v.2 system
Prognostic factor- 2 | 12 months follow up
  Survival rate
Prognostic factor- 1 | 24 months follow up
  Surgery-related adverse events collected by SAVES-v.2 system
Prognostic factor- 2 | 24 months follow up
  Survival rate
Prognostic factor- 1 | 36 months follow up
  Surgery-related adverse events collected by SAVES-v.2 system
Prognostic factor- 2 | 36 months follow up
  Survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Terzi, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided